CLINICAL TRIAL: NCT06477302
Title: Construction and Psychometric Properties of the Therapeutic Adherence Scale for Respiratory Rehabilitation in Lung Cancer (STA-RR-LC).
Brief Title: Scale of Therapeutic Adherence to Respiratory Rahabilitation for Lung Cancer
Acronym: STA-RR-LC
Status: Recruiting | Type: Observational
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Oscar Gerardo Arrieta Rodríguez, Dr., Instituto Nacional de Cancerologia de Mexico
Other Study IDs: (023/039/ICI)(CEI/045/23)
Record Dates: First submitted 2024-06-21; First posted 2024-06-27 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer
Keywords: pulmonary rehabilitation; therapeutic adherence; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adherence group: Patients with a confirmed diagnosis of lung cancer who are undergoing respiratory rehabilitation treatment with at least one month of monitoring and follow-up.
  Interventions: Behavioral: Scale of Therapeutic Adherence to Respiratory Rahabilitation for Lung Cancer (STA-RR-LC)

INTERVENTIONS:
Behavioral: Scale of Therapeutic Adherence to Respiratory Rahabilitation for Lung Cancer (STA-RR-LC) — Patients will be given a measurement instrument to determine the level of therapeutic adherence.

SUMMARY:
The goal of this non experimental, transversal instrument study is to Construct and determine the reliability and validity of the Scale of Therapeutic Adherence for Respiratory Rehabilitation in Lung Cancer in Mexican patients with a lung cancer diagnosis.

The main question it aims to answer is: What is the reliability and validity of the Scale of Therapeutic Adherence for Respiratory Rehabilitation in Lung Cancer of the patients with this diagnosis that are currently undergoing an assessment or follow up program of Respiratory Rehabilitation?

The Scale of Therapeutic Adherence for Respiratory Rehabilitation in Lung Cancer (STA-RR-LC) will be psychometrically valid and reliable for the evaluation of therapeutic adherence on patients with lung cancer that are undergoing an assessment or follow up of Respiratory Rehabilitation.Participants will be asked to fill out an Identification card and fill out the fifty-six items presented on the STA-RR-LC.

DETAILED DESCRIPTION:
For the recruitment patients with lung cancer diagnosis that arrive at the Respiratory Rehabilitation service will be asked if they are willing to participate and fill out the STA.

It will be explained to them as clearly as possible the objective, procedure, risks and benefits of the study and a copy of the Informed Consent will be provided. Lung cancer patients attending the Pulmonary Rehabilitation service will be approached and a verbal explanation of the study will be given.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with lung cancer (SCLC and NSCLC).
* Over 18 years of age.
* Voluntary participation by understanding and accepting the informed consent letter.
* Patients undergoing Respiratory Rehabilitation treatment with one month assessment and follow-up.
* Patients in active medical treatment.
* Any clinical stage.
* Karnofsky Index ≥ 70.

Exclusion Criteria:

* Severe hearing or visual problems that prevent them from understanding the instructions and answering the instruments (this will be identified as reported in the clinical record file).
* Severe psychiatric conditions (schizophrenia or psychotic disorders) and/or addiction to any psychoactive substance (this will be identified as reported in the INCanet file).
* Attentional or memory problems that prevent them from understanding the instructions and answering the instruments (this will be identified as reported in the INCanet file).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient registered in the national cancer center with respiratory rehabilitation follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 281 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2026-06-23 (Estimated); Study Completion 2027-06-23 (Estimated)

PRIMARY OUTCOMES:
Contruction of the Scale of Therapeutic Adherence for Respiratory Rehabilitation in Lung Cancer (STA-RR-LC) | the STA-RR-LC will be applied for one time and as soon as the patient has completed one month attending the Respiratory Rehabilitation Service.
  The validity of the construction is carried out with an exploratory factor analysis using the Maximum Likelihood extraction method and the oblique rotation (direct Oblimin). Confiability is determitated using the Alpha of Cronbach coefficient.

SECONDARY OUTCOMES:
Verify the concurrent validity of the instrument | the STA-RR-LC will be applied one time, as soon as the patient has completed one month attending the Respiratory Rehabilitation Service
  It will be verified using the current scores of the European Organisation for Research and Treatment of Cancer, specifically the Module of Lung Cancer (EORTC-QLQ-LC29).

CONTACTS AND LOCATIONS:
Overall Officials: Oscar G Arrieta, MD, Principal Investigator — Instituto Nacional de Cancerologia (INCan) Mexico
Locations (1):
- Instituto Nacional de Cancerologia, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] McFarland DC, Jutagir DR, Miller A, Nelson C. Physical problem list accompanying the distress thermometer: Its associations with psychological symptoms and survival in patients with metastatic lung cancer. Psychooncology. 2020 May;29(5):910-919. doi: 10.1002/pon.5367. Epub 2020 Mar 11. PMID 32096582
- [Background] Eggen AC, Reyners AKL, Shen G, Bosma I, Jalving M, Leighl NB, Liu G, Richard NM, Mah K, Shultz DB, Edelstein K, Rodin G. Death Anxiety in Patients With Metastatic Non-Small Cell Lung Cancer With and Without Brain Metastases. J Pain Symptom Manage. 2020 Aug;60(2):422-429.e1. doi: 10.1016/j.jpainsymman.2020.02.023. Epub 2020 Mar 5. PMID 32145337
- [Background] Tan H, Chen S, Ercolano E, Lazenby M, Davies M, Chen J, McCorkle R. The prevalence and related factors associated with psychosocial distress among 420 hospitalised lung cancer patients in China: A case study. Eur J Cancer Care (Engl). 2019 Jul;28(4):e13046. doi: 10.1111/ecc.13046. Epub 2019 Apr 24. PMID 31016811
- [Background] Papadopoulos D, Kiagia M, Charpidou A, Gkiozos I, Syrigos K. Psychological correlates of sleep quality in lung cancer patients under chemotherapy: A single-center cross-sectional study. Psychooncology. 2019 Sep;28(9):1879-1886. doi: 10.1002/pon.5167. Epub 2019 Jul 18. PMID 31264308
- [Background] Ernst J, Mehnert A, Dietz A, Hornemann B, Esser P. Perceived stigmatization and its impact on quality of life - results from a large register-based study including breast, colon, prostate and lung cancer patients. BMC Cancer. 2017 Nov 9;17(1):741. doi: 10.1186/s12885-017-3742-2. PMID 29121876
- [Background] Vodermaier A, Lucas S, Linden W, Olson R. Anxiety After Diagnosis Predicts Lung Cancer-Specific and Overall Survival in Patients With Stage III Non-Small Cell Lung Cancer: A Population-Based Cohort Study. J Pain Symptom Manage. 2017 Jun;53(6):1057-1065. doi: 10.1016/j.jpainsymman.2016.12.338. Epub 2017 Jan 4. PMID 28063862
- [Background] Arrieta O, Angulo LP, Nunez-Valencia C, Dorantes-Gallareta Y, Macedo EO, Martinez-Lopez D, Alvarado S, Corona-Cruz JF, Onate-Ocana LF. Association of depression and anxiety on quality of life, treatment adherence, and prognosis in patients with advanced non-small cell lung cancer. Ann Surg Oncol. 2013 Jun;20(6):1941-8. doi: 10.1245/s10434-012-2793-5. Epub 2012 Dec 22. PMID 23263699
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Saad FA, Busque C, Vitiello L, Danieli GA. DXS997 localized to intron 48 of dystrophin. Hum Mol Genet. 1994 Jun;3(6):1034. doi: 10.1093/hmg/3.6.1033. No abstract available. PMID 7951226